CLINICAL TRIAL: NCT05048147
Title: Community Mobilization for Improved Clean Cookstove Uptake, Household Air Pollution Reduction, and Hypertension Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-00586; R01HL157091 (NIH)
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Hypertension; Cardiovascular diseases; Clean cookstove; Clean fuel; Community mobilization; Household air pollution
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM Intervention Group (Experimental): Cluster. RCT of 16 urban and rural communities. Community mobilizers and health education officers will facilitate use of CF-CS (bioethanol and LPG fuels/stoves) and educate households on HAP exposure throughout the intervention period
  Interventions: Behavioral: Community Mobilization
- Self-Directed Group (No Intervention): Receive information on CFCS use and education on HAP in 16 urban and rural communities; will not receive the CM intervention

INTERVENTIONS:
Behavioral: Community Mobilization — The Community Mobilization (CM) strategy will include: (1) Community advisory board [comprising local community-based organizations, government officials, and residents], that will provide leadership support and buy-in for adoption of Clean Fuel- Clean- Stove (CF-CS) use; (2) Trained MoH community health extension workers, community health officers, community mobilizers and health education officers, who will form community action teams (CAT) to facilitate the implementation of CF-CS use via provision of support, knowledge exchange and performance feedback to the primary cooks in participating households; (3) Community dialogues with residents and households focused on shared concerns on the significance and importance of CF-CS use.
  Arms: CM Intervention Group

SUMMARY:
Using a focused implementation research framework, the EPIS (Exploration, Preparation, Implementation and Sustainment) model in a type-2 hybrid design, the study will be conducted in 3 phases: 1) A pre-implementation phase that will use the Exploration and Preparation domains of EPIS to: a) explore barriers and facilitators of Clean Fuel- Clean- Stove (CF-CS) use, and b) develop a culturally-tailored CM strategy for CF-CS use; 2) An Implementation phase that will use the Implementation domain of EPIS to compare in a cluster RCT of 32 peri-urban communities (640 households), the effect of CM vs. a self-directed condition (i.e. receipt of information on CF-CS use without CM) on adoption of CF-CS use; and systolic BP reduction; 3) A post-implementation phase that will use the Sustainment domain of EPIS to evaluate the effect of CM strategy vs. self-directed condition on sustainability of the CF-CS use in 640 households across the randomly assigned 32 peri-urban communities in Nigeria. The Lagos State University College of Medicine (LASUCOM) working with the MOH will oversee research coordination in Nigeria.

DETAILED DESCRIPTION:
This study will use CM to engage in the community dialogues, organize outreach facilitation, and advocacy for the adoption of bioethanol-based and liquified petroleum gas (LPG) CF-CS across participating households. The choice of CM strategy is deliberate because, unlike western culture, African cultures are largely based on communal hierarchy.

ELIGIBILITY:
Inclusion Criteria:

* Primary adult must be a female cook;
* Must not have a paid housemaid;
* Family size must be a minimum of 2 and no more than 7 members;
* Family must use Kerosene, charcoal, LPG, or firewood as primary cooking fuel;
* The person spoken to at enrollment must be the home key decision maker;
* Must have no plans for relocation in the next year.

Exclusion Criteria:

• Does not meet the inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants who have Adopted CF-CS at Baseline | Baseline
  Adoption defined as utilization of the CF-CS for more than 50% of cooking activities based on the metric developed by the Global Alliance for Clean Cookstoves. All traditional stoves and the bioethanol-based CF-CS in the participating households will be equipped with the iButtons SUMs to assess their use. Trained study staff will collect iButton temperature data during household visits.
Percent of Participants who have Adopted CF-CS at Month 12 | Month 12
  Adoption defined as utilization of the CF-CS for more than 50% of cooking activities based on the metric developed by the Global Alliance for Clean Cookstoves. All traditional stoves and the bioethanol-based CF-CS in the participating households will be equipped with the iButtons SUMs to assess their use. Trained study staff will collect iButton temperature data during household visits.

SECONDARY OUTCOMES:
Change in Mean Systolic Blood Pressure from Baseline to Month 12 | Baseline, Month 12
  Blood pressure readings assessed with a validated automated BP device. At each visit, three readings will be taken by trained research coordinators using an automated BP monitor. The average of three BP readings will be used as the measure for each study visit.
Percent of Participants who Have Adopted CF-CS at Month 24 | Month 24
  Measure of sustainability. Adoption defined as utilization of the CF-CS for more than 50% of cooking activities based on the metric developed by the Global Alliance for Clean Cookstoves. All traditional stoves and the bioethanol-based CF-CS in the participating households will be equipped with the iButtons SUMs to assess their use. Trained study staff will collect iButton temperature data during household visits.

CONTACTS AND LOCATIONS:
Overall Officials: Olugbenga Ogedegbe, MD, Principal Investigator — NYU Langone Health; Christopher O Olopade, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. To achieve aims in the approved proposal. Requests should be directed to olugbenga.ogedegbe@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Onakomaiya DO, Mishra S, Colvin C, Ogunyemi R, Aderibigbe AA, Fagbemi T, Adeniji MR, Li S, Kanneh N, Aifah A, Vedanthan R, Olopade CO, Wright K, Ogedegbe G, Wall SP. Stakeholders' perspectives on implementation of a clean fuel: clean stove intervention for reduction of household air pollution and hypertension in Lagos, Nigeria - a qualitative study. BMJ Open. 2026 Jan 9;16(1):e101218. doi: 10.1136/bmjopen-2025-101218. PMID 41513415
- [Derived] Wright O, Olopade CO, Aifah AA, Fagbemi T, Hade EM, Mishra S, Onakomaiya DO, Kanneh N, Chen W, Colvin CL, Ogunyemi R, Sogbossi E, Erinosho E, Ojengbede O, Taiwo O, Johnson MA, Vedanthan R, Wall S, Lwelunmor J, Idris O, Ogedegbe G. Community mobilisation for adoption of clean cookstoves and clean fuel to reduce household air pollution and blood pressure in Lagos, Nigeria: protocol for a cluster-randomised trial. BMJ Open. 2025 Sep 10;15(9):e098483. doi: 10.1136/bmjopen-2024-098483. PMID 40935430

DOCUMENTS (1):
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT05048147/ICF_000.pdf